CLINICAL TRIAL: NCT07295600
Title: Postprandial Effect of Isocaloric Challenge Meals Enriched With Indigenous Fruits and Vegetables on Glucose Metabolism in Individuals With Type 2 Diabetes in Wakiso District, Uganda
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Christophe Matthys, Proffessor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Postprandial studies
Record Dates: First submitted 2025-12-03; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes; Cardiometabolic Health
Keywords: Type 2 diabetes; Challenge meals; Postprandial; Glucose metabolism; Indigenous fruits and Vegetables
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vegetables

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Challenge meal enriched with Hibiscus sabdariffa (Hibiscus) (Experimental)
  Interventions: Other: Indigenous Fruit and vegetable.
- Challenge meal enriched with Solunum anguivi (Forest bitter berries) (Experimental)
  Interventions: Other: Indigenous Fruit and vegetable.
- Challenge meal enriched withTamarindus indica (Tamarind) (Experimental)
  Interventions: Other: Indigenous Fruit and vegetable.
- Reference meal one (Active Comparator)
  Interventions: Other: Challenge meal that resembles the oral glucose tolerance test.
- Reference meal two (Active Comparator)
  Interventions: Other: Challenge meal that resembles the oral glucose tolerance test.

INTERVENTIONS:
Other: Indigenous Fruit and vegetable. — Indigenous fruit and vegetable freeze dried powder.
  Arms: Challenge meal enriched with Hibiscus sabdariffa (Hibiscus); Challenge meal enriched with Solunum anguivi (Forest bitter berries); Challenge meal enriched withTamarindus indica (Tamarind)
Other: Challenge meal that resembles the oral glucose tolerance test. — Isocaloric challenge meal
  Arms: Reference meal one; Reference meal two

SUMMARY:
The goal of this clinical trial is to evaluate changes in glucose and lipid levels after consuming challenge meals enriched with selected indigenous fruits and vegetables in people living with type 2 diabetes in Wakiso district.

The main question to answer is:

Does the consumption of challenge meals enriched with indigenous fruits and vegetables improve glucose and lipid levels among people living with type 2 diabetes? Researchers will compare the effects of different challenge meals on glucose and lipid levels to identify the indigenous fruit and vegetable with the strongest glucose- and lipid-lowering effects.

Participants will:

Consume five challenge meals over 5 weeks. Visit the study site after a 5-7 day rest period to consume the challenge meal and complete the tests.

DETAILED DESCRIPTION:
In a postprandial study, cardiometabolic health outcomes will be assessed on each 3-hour test day, comprising the consumption of one challenge meal enriched with any of the three indigenous fruits and vegetable based powders. The study participants will be randomly allocated to consume one challenge meal enriched with one of the three indigenous fruits and vegetable based powders on each study day. The indigenous fruits and vegetable based powders will contain a dose of 760 mg of total polyphenol. The three indigenous fruits and vegetable will include: Hibiscus sabdariffa (Hibiscus), Solunum anguivi (Forest bitter berries), and Tamarindus indica (Tamarind). There will be an additional two reference challenge meals administered to determine within-subject variability. A 5 to 7-day washout period will be observed between each postprandial study to prevent any carryover effect. The participants in the study will not be informed of the ingredients in the challenge meals. The total study duration will be 5 weeks. Measurements will be performed on each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood sugar >= [7 mmol/L](based on medical records)
* Diabetic regimen for at least 6 months
* Type 2 diabetes
* Plans to continue staying in the same location for the next 6 months

Exclusion Criteria:

* Taking dietary supplements
* Type 1 diabetes
* Tuberculosis co-infection
* Renal failure
* Liver cirrhosis
* Chronic pancreatitis
* Pregnancy and Lactation
* Regular sports activity
* Parallel participation in another clinical trial
* On treatment for dyslipidaemia,
* On treatment for hypertension
* Very low blood pressure (< 90/50 mmHg)
* Allergic reactions to test products

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incremental area under the curve blood glucose | From enrollment at each of the five postprandial visits, until the end of the postprandial study which will last five weeks
  Blood glucose analysis for blood samples collected at 8 different time points:0, 15, 30, 60, 90, 120, 150 and 180 minutes

SECONDARY OUTCOMES:
Incremental area under the curve blood triglyceride | From enrollment at each of the five postprandial visits, until the end of the postprandial study which will last five weeks
  Blood Triglyceride analysis for blood samples collected at 8 different time points:0, 15, 30, 60, 90, 120, 150 and 180 minutes
Incremental area under the curve high density lipoprotein cholestrol (HDL) | From enrollment at each of the five postprandial visits, until the end of the postprandial study which will last five weeks
  Blood HDL analysis for blood samples collected at 8 different time points:0, 15, 30, 60, 90, 120, 150 and 180 minutes
Incremental area under the curve low density lipoprotein cholestrol (LDL) | From enrollment at each of the five postprandial visits, until the end of the postprandial study which will last five weeks
  Blood LDL analysis for blood samples collected at 8 different time points:0, 15, 30, 60, 90, 120, 150 and 180 minutes
Incremental area under the curve total cholestrol | From enrollment at each of the five postprandial visits, until the end of the postprandial study which will last five weeks
  Blood cholestrol analysis for blood samples collected at 8 different time points:0, 15, 30, 60, 90, 120, 150 and 180 minutes
Incremental area under the curve plasma polyphenol metabolites | From enrollment at each of the five postprandial visits, until the end of the postprandial study which will last five weeks
  Plasma polyphenol metabolite analysis for blood samples collected at 8 different time points:0, 15, 30, 60, 90, 120, 150 and 180 minutes

OTHER OUTCOMES:
Body mass Index (BMI) | BMI will be calculated only on day one of the study that lasts five weeks
  BMI will be calculated using height and weight
Fat mass | Fat mass will be calculated only on day one of the study that lasts five weeks
  Bioelectrical impedence analysis will be performed
Waist circumference | Waist circumference will be calculated only on day one of the study that lasts five weeks
  Wait circumference will be measured using a measuring tape

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Matthys, Phd, Principal Investigator — KU Leuven University, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) Sharing Statement Plan to Share IPD:
  Plan Description: All the data generated during this study will comply with the prevailing standards and guidelines in documenting and depositing data sets.
  The results from this research will be disseminated in presentations at public lectures, scientific institutions and meetings, and/or publication in reputable journals. Data sharing will be performed in compliance with the International Committee of Medical Journal Editors. Individual de-identified participant data will be shared. In particular, individual participant data that underlie the results reported in our articles, after de-identification (text, tables, figures and appendices).
  Supporting Materials: Study Protocol Informed Consent Form (ICF) Analytic Code Time Frame: Data will become available from 9-36 months after the publication of the study results by the research team.
  Access Criteria: Data will only be shared with investigators
Supporting Information: Study Protocol, SAP
Time Frame: 9 to 18 months after article publication.